CLINICAL TRIAL: NCT04931706
Title: Double Magnetic-assisted Single-port Nissen Sleeve
Brief Title: Nissen Sleeve by Single Port With Magnetic Assistance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unidad Internacional de Cirugia Bariatrica y Metabolica (Other)
Responsible Party: Principal Investigator, Guillermo Borjas, Director, Unidad Internacional de Cirugia Bariatrica y Metabolica
Other Study IDs: UICBM
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Bariatric Surgery Candidate; Obesity; GERD
Keywords: Bariatric Surgery; Magnetic assisted; Singe port; Nissen Sleeve
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- N-Sleve patients: Patient that were selected for surgery
  Interventions: Other: Magnetics Assisted by Singe port

INTERVENTIONS:
Other: Magnetics Assisted by Singe port — Use of magnet for assistance through the surgery, and a novel approach as it is single port

SUMMARY:
New approach for Nissen Sleeve Gastrectomy by single port using double magnetic system

DETAILED DESCRIPTION:
A bariatric surgery is performed for weight loss and esophagogastric reflux, called Nissen Sleeve, in which a new approach is used which is the only port that helps to shorten the hospital stay because it decreases postoperative pain as well as increases the esthetic Ad benefit. In addition, a system of magnets is used to assist in different steps of the surgery for the correct retraction of the tissues and to be able to suture or perform the correct dissection.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with controlled comorbidities suffering from obesity and GERD.

Exclusion Criteria:

* Patients with pacemakers, psychiatric problems or uncontrolled metabolic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the UICBM from Venezuela-Colombia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-05 (Actual); Primary Completion 2023-06-05 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Surgical Complications | 1 month
  any adverse event during the surgery
Surgical time | 30 minutes
  how long does the surgery take
Weight loss follow up | 1 month
  Kg that the patient loss

CONTACTS AND LOCATIONS:
Overall Officials: Andres Maldonado, M.D., Principal Investigator — UICBM
Locations (1):
- Unidad Internacional de Cirugia Bariatric y Metabolica, Maracaibo, Zulia, Venezuela

IPD SHARING:
Plan to Share IPD: Undecided